CLINICAL TRIAL: NCT05700838
Title: Refining Cough Skill Training in Parkinson's Disease and Dysphagia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Principal Investigator, Michelle Troche, Associate Professor, Lab Director, Teachers College, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-016
Record Dates: First submitted 2022-12-21; First posted 2023-01-26 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease; Dysphagia
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cough Skill Training (Experimental): During cough skill training, participants will be seated in front of a computer with real-time visualization of their cough waveform. A target line will be provided, and participants will be instructed to perform a single voluntary cough so that their peak flow is within the target's range. Participants will be instructed to continue the cough training regardless of initial accuracy.
  Interventions: Behavioral: Cough Skill Training - with Variable Practice

INTERVENTIONS:
Behavioral: Cough Skill Training - with Variable Practice — Variable practice will involve three targets that reflect a range of cough airflows, including "strong", "moderate", and "weak" coughs.

SUMMARY:
Airway protection deficits (cough and swallowing) are prevalent and pervasive in Parkinson's disease (PD), contributing to adverse health outcomes like pneumonia. This study aims to refine cough skill training by examining whether variable versus constant practice conditions improve cough outcomes in people with PD. In addition, this study will provide insight into optimal respiratory adaptations that occur during training to support cough effectiveness, resulting in immediately translatable treatments to improve airway protection-related health outcomes in people with neurodegenerative disease.

ELIGIBILITY:
Inclusion criteria:

* 40 years of age or older
* have dysphagia as documented by a penetration-aspiration score > 2 on a flexible endoscopic evaluation of swallowing
* have cough disorder as defined as a maximal voluntary cough peak flow < 5 L/s
* have no history of other neurological disorders, head and neck cancer, respiratory disease, smoking within 5 years, uncontrolled hypertension, or allergy to capsaicin (reflex cough stimulus)

Exclusion criteria:

* unable to participate due to neuropsychological dysfunction (i.e., dementia with a score of < 19 on the Montreal Cognitive Assessment)
* actively participating in other cough or swallowing treatments

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Change in Peak Expiratory Flow Rate | Before to after two sessions of cough variable practice training over two weeks
  Cough Strength

SECONDARY OUTCOMES:
Change in Respiratory Kinematics, specifically lung volume excursion | Before to after two sessions of cough variable practice training over two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No